CLINICAL TRIAL: NCT00142415
Title: Phase I/II Study of Increasing Doses of Lutetium-177 Labeled Chimeric Monoclonal Antibody cG250 (177^Lu-DOTA-cG250) in Patients With Advanced Renal Cancer
Brief Title: Phase I/II Dose-escalation Study of Lutetium-177-labeled cG250 in Patients With Advanced Renal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2003-006
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Advanced Renal Cell Carcinoma; Clear Cell Renal Cell Carcinoma (CCRCC); Lutetium-177; 177-Lu; cG250; DOTA-cG250; Monoclonal Antibody
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 (Experimental): Subjects received an initial single dose of 10 mg of cG250 coupled to DOTA and labeled with 30 mCi/m^2 of 177-Lu.
  Interventions: Drug: 111-In-DOTA-cG250; Drug: 177-Lu-DOTA-cG250
- Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 (Experimental): Subjects received an initial single dose of 10 mg of cG250 coupled to DOTA and labeled with 40 mCi/m^2 of 177-Lu.
  Interventions: Drug: 111-In-DOTA-cG250; Drug: 177-Lu-DOTA-cG250
- Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 (Experimental): Subjects received an initial single dose of 10 mg of cG250 coupled to DOTA and labeled with 50 mCi/m^2 of 177-Lu.
  Interventions: Drug: 111-In-DOTA-cG250; Drug: 177-Lu-DOTA-cG250
- Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 (Experimental): Subjects received an initial single dose of 10 mg of cG250 coupled to DOTA and labeled with 60 mCi/m^2 of 177-Lu.
  Interventions: Drug: 111-In-DOTA-cG250; Drug: 177-Lu-DOTA-cG250
- Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 (Experimental): Subjects received an initial single dose of 10 mg of cG250 coupled to DOTA and labeled with 70 mCi/m^2 of 177-Lu.
  Interventions: Drug: 111-In-DOTA-cG250; Drug: 177-Lu-DOTA-cG250
- Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250 (Experimental): Subjects received an initial single dose of 10 mg of cG250 coupled to DOTA and labeled with 65 mCi/m^2 of 177-Lu.
  Interventions: Drug: 111-In-DOTA-cG250; Drug: 177-Lu-DOTA-cG250

INTERVENTIONS:
Drug: 111-In-DOTA-cG250 — On Day 1, each subject received a single intravenous (IV) infusion of 10 mg of cG250 coupled to DOTA and labeled with 5 mCi of 111-In.
  Other Names: cG250; DOTA-cG250; cG250-In111
Drug: 177-Lu-DOTA-cG250 — On Day 8, 9, or 10, each subject received a single IV infusion of 10 mg of cG250 coupled to DOTA and labeled with a dose of 177-Lu at a starting dose of 30 mCi/m^2 in the initial cohort.
  Other Names: cG250; DOTA-cG250; cG200-Lu177

SUMMARY:
This was a Phase I/II, single-center, dose-escalation study. 177-Lutetium-1,4,7,10-tetraazacyclododecane-1,4,7,10-tetraacetic acid-cG250 (177-Lu-DOTA-cG250) was administered at a starting dose of 30 mCi/m^2 of 177-Lu (fixed dose of 10 mg cG250) and escalated in increments of 10 mCi/m^2 of 177-Lu in sequentially enrolled cohorts according to a standard 3 + 3 design until determination of the maximum tolerated dose (MTD). The primary objectives were to determine the safety, targeting, and dosimetry of 177-Lu-DOTA-cG250 in subjects with advanced renal cell carcinoma. The secondary objective was measurement of tumor response according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0.

DETAILED DESCRIPTION:
Prior to administration of 177-Lu-DOTA-cG250, subjects received 5 mCi/10 mg of the 111-Indium-DOTA-cG250 (111-In-DOTA-cG250) antibody (an imaging dose). Whole body and blood measurements of radioactivity were obtained on at least 3 occasions for 1 week to determine targeting and dosimetry. If at least one known and evaluable metastatic lesion was visualized with 111-In-DOTA-cG250, a single dose of therapeutic 177-Lu-DOTA-cG250 was administered the following week. In the absence of disease progression and after recovery from toxicity, subjects may have been retreated no sooner than 12 weeks after the previous treatment with a dose of no more than 75% of the previous dose, for a total of not more than 3 treatments. Only subjects with normal pharmacokinetics on the diagnostic 111-In-DOTA-cG250 study (indicative of human anti-chimeric antibody [HACA] negativity) were eligible for re-treatment.

Subjects in the initial cohort were enrolled sequentially to receive 30 mCi/m^2 of 177-Lu-DOTA-cG250 (fixed dose of 10 mg cG250). In the absence of a dose-limiting toxicity, the dose was escalated in each subsequent cohort in 10 mCi/m^2 increments of 177-Lu. At least 3 subjects per dose level were followed for up to 12 weeks with imaging, biochemical, and hematologic tests. Safety was monitored continuously throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with proven advanced and progressive renal cell carcinoma (RCC) of the clear cell type.
2. At least one evaluable lesion < 5 cm.
3. Karnofsky performance status ≥ 70%.
4. Laboratory values obtained < 14 days prior to registration:

   * White blood cells (WBC) ≥ 3.5 × 10^9/L
   * Platelet count ≥ 100 × 10^9/L
   * Hemoglobin ≥ 6 mmol/L
   * Total bilirubin ≤ 2 × upper limit of normal (ULN)
   * Aspartate aminotransferase and alanine aminotransferase ≤ 3 × ULN (< 5 × ULN if liver metastases present)
   * Serum creatinine ≤ 2 × ULN
5. Negative pregnancy test for women of childbearing potential (urine or serum).
6. Age over 18 years.
7. Ability to provide written informed consent.

Exclusion Criteria:

1. Known metastases to the brain.
2. Untreated hypercalcemia.
3. Metastatic disease limited to the bone.
4. Pre-exposure to murine/chimeric antibody therapy.
5. Chemotherapy, external beam radiation or immunotherapy within 4 weeks prior to study. Limited field external beam radiotherapy to prevent pathological fractures was allowed, when unirradiated, evaluable lesions were present elsewhere.
6. Cardiac disease with New York Heart Association classification of III or IV.
7. Subjects who were pregnant, nursing or of reproductive potential and were not practicing an effective method of contraception.
8. Any unrelated illness, e.g., active infection, inflammation, medical condition or laboratory abnormality, that in the judgement of the investigator would have significantly affected the subject's clinical status.
9. Life expectancy < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W.J.G. Oyen, MD, Principal Investigator — Department of Nuclear Medicine, University Medical Center Nijmegen; P.F.A. Mulders, MD, Principal Investigator — Department of Urology, University Medical Center Nijmegen
Locations (1):
- University Medical Center Nijmegen, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data have been published

REFERENCES:
- [Result] Stillebroer AB, Boerman OC, Desar IM, Boers-Sonderen MJ, van Herpen CM, Langenhuijsen JF, Smith-Jones PM, Oosterwijk E, Oyen WJ, Mulders PF. Phase 1 radioimmunotherapy study with lutetium 177-labeled anti-carbonic anhydrase IX monoclonal antibody girentuximab in patients with advanced renal cell carcinoma. Eur Urol. 2013 Sep;64(3):478-85. doi: 10.1016/j.eururo.2012.08.024. Epub 2012 Aug 21. PMID 22980441
- [Result] Stillebroer AB, Zegers CM, Boerman OC, Oosterwijk E, Mulders PF, O'Donoghue JA, Visser EP, Oyen WJ. Dosimetric analysis of 177Lu-cG250 radioimmunotherapy in renal cell carcinoma patients: correlation with myelotoxicity and pretherapeutic absorbed dose predictions based on 111In-cG250 imaging. J Nucl Med. 2012 Jan;53(1):82-9. doi: 10.2967/jnumed.111.094896. Epub 2011 Dec 12. PMID 22159179
- See also: Stillebroer et al. J Nucl Med 2012; 53(1):82-89 — http://jnm.snmjournals.org/content/53/1/82.long

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250: 111-In-DOTA-cG250: On Day 1, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 5 mCi of 111-In.
  177-Lu-DOTA-cG250: On Day 8, 9, or 10, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 30 mCi/m^2 of 177-Lu.
- Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250: 111-In-DOTA-cG250: On Day 1, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 5 mCi of 111-In.
  177-Lu-DOTA-cG250: On Day 8, 9, or 10, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 40 mCi/m^2 of 177-Lu.
- Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250: 111-In-DOTA-cG250: On Day 1, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 5 mCi of 111-In.
  177-Lu-DOTA-cG250: On Day 8, 9, or 10, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 50 mCi/m^2 of 177-Lu.
- Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250: 111-In-DOTA-cG250: On Day 1, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 5 mCi of 111-In.
  177-Lu-DOTA-cG250: On Day 8, 9, or 10, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 60 mCi/m^2 of 177-Lu.
- Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250: 111-In-DOTA-cG250: On Day 1, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 5 mCi of 111-In.
  177-Lu-DOTA-cG250: On Day 8, 9, or 10, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 70 mCi/m^2 of 177-Lu.
- Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250: 111-In-DOTA-cG250: On Day 1, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 5 mCi of 111-In.
  177-Lu-DOTA-cG250: On Day 8, 9, or 10, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 65 mCi/m^2 of 177-Lu.
Period: Overall Study
Arm/Group | Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250
Started | 3 | 3 | 6 | 3 | 3 | 8
Completed (Defined as completion of Cycle 1 (ie, received 111-In-DOTA-cG250 and 177-Lu-DOTA-cG250)) | 3 | 3 | 6 | 3 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set comprises all subjects who received at least 1 dose of 111-In-DOTA-cG250 or 177-Lu-DOTA-cG250.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3 | 8 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.74) | 60.7 (12.86) | 64.7 (7.87) | 51.3 (6.11) | 44.7 (13.80) | 58.3 (8.94) | 57.8 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 0 | 1 | 1 | 5
  Male | 1 | 3 | 5 | 3 | 2 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 3 | 6 | 3 | 3 | 6 | 21
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 0 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 6 | 3 | 3 | 8 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 3 | 3 | 6 | 3 | 3 | 8 | 26
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.0 (1.29) | 28.6 (3.38) | 27.2 (4.52) | 28.5 (5.84) | 31.2 (5.35) | 26.7 (1.78) | 27.3 (3.95)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Description: Toxicity was graded in accordance with the NCI CTCAE version 3.0. Treatment-emergent adverse events (TEAEs) were reported based on clinical laboratory tests, physical examinations, and vital signs from pre-treatment through 4 weeks after the last dose of study treatment.
Time Frame: Up to 1 year
Population: The Safety Analysis Set comprises all subjects who received at least 1 dose of 111-In-DOTA-cG250 or 177-Lu-DOTA-cG250.
Measure: Number; unit: participants
Arm/Group | Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3 | 8
participants
  Any TEAE | 3 | 3 | 6 | 3 | 2 | 6
  Maximum Grade 3 TEAE | 0 | 0 | 1 | 0 | 0 | 3
  Maximum Grade 4 TEAE | 0 | 1 | 1 | 0 | 2 | 2
  Treatment-related TEAE | 2 | 3 | 6 | 3 | 2 | 6
  SAE | 0 | 2 | 1 | 0 | 1 | 2
  Death | 0 | 0 | 1 | 0 | 0 | 0
  TEAE Leading to Discontinuation | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Dose-limiting Toxicity (DLT) During Cycle 1
Description: Subjects were monitored for AEs for ≥ 8 weeks after the last infusion of 177-Lu-DOTA-cG250 before dose escalation could be implemented. Toxicity was graded in accordance with the NCI CTCAE version 3.0. DLT was defined as the following treatment-related events: ≥ Grade 3 non-hematologic toxicity; ≥ Grade 4 hematologic toxicity (platelets < 25 × 10^9/L or leukocytes < 1.0 × 10^9/L) that persisted for > 4 weeks except anemia; thrombocytopenia < 10 × 10^9/L; clinically relevant myelotoxicity that required hospitalization and/or blood product transfusion (e.g., uncontrolled bleeding, infections that had to be treated clinically).
Time Frame: 12 weeks
Population: The Safety Analysis Set comprises all subjects who received at least 1 dose of 111-In-DOTA-cG250 or 177-Lu-DOTA-cG250.
Measure: Number; unit: participants
Arm/Group | Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 3 | 8
participants
  Any DLT | 0 | 0 | 1 | 0 | 2 | 1
  Grade 4 Thrombocytopenia | 0 | 0 | 1 | 0 | 2 | 1
  Grade 4 Leukopenia | 0 | 0 | 0 | 0 | 2 | 0
  Grade 4 Neutropenia | 0 | 0 | 1 | 0 | 0 | 1
  Grade 3 Epistaxis | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Fatigue | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Hematoma | 0 | 0 | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 vs Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 vs Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 vs Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 vs Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 vs Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250; Test type: Other — The maximum tolerated dose (MTD) was determined using a standard 3 + 3 dose-escalation design. The occurrence of DLTs was compared across cohorts; Maximum tolerated dose (mCi/m^2) = 65

3. Primary Outcome: Radiation Absorbed Doses by Organ for 177-Lu-cG250
Description: After each 177-Lu-cG250 administration, 3 whole-body scintigrams were acquired (directly after injection and 2-4 days and 5-7 days post-injection) and blood samples were drawn at 5, 30, 60, and 120 min, 2-4 days, and 5-7 days post-infusion. Estimated radiation absorbed doses were calculated according to the Medical Internal Radiation Dose scheme, which permits estimation of the factors required to calculate dose to one organ attributable to a source in another organ.
Time Frame: 12 weeks
Population: The Dosimetry Evaluable Analysis Set comprises all subjects who received at least 1 dose of 177-Lu-cG250.
Measure: Mean (Standard Deviation); unit: mGy/MBq
Groups:
- Dosimetry Evaluable Analysis Set: 111-In-DOTA-cG250: On Day 1, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 5 mCi of 111-In.
  177-Lu-DOTA-cG250: On Day 8, 9, or 10, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 30 to 70 mCi/m^2 of 177-Lu.
Arm/Group | Dosimetry Evaluable Analysis Set
Number analyzed (Participants) | 20
mGy/MBq
  Whole Body | 0.24 (0.04)
  Liver | 1.26 (0.25)
  Heart Wall | 0.76 (0.16)
  Red Marrow (Image-based) | 0.44 (0.07)
  Red Marrow (Blood-based) | 0.35 (0.07)
  Kidney | 1.30 (0.35)
  Lungs | 0.49 (0.13)
  Testes | 1.90 (0.45)
  Metastases | 5.72 (4.52)

4. Secondary Outcome: Number of Subjects With Best Overall Tumor Response
Description: Tumor responses were evaluated using computed tomography and categorized according to RECIST v1.0 at baseline and at the end of every cycle (every 12 weeks) or after recovery from toxicity. Per RECIST v1.0 for target lesions and assessed by MRI: Complete Response (CR): Disappearance of all target lesions [no evidence of disease]; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 9 months
Population: The Evaluable Analysis Set comprises subjects who completed Cycle 1 (ie, received both 111-In-DOTA-cG250 and 177-Lu-DOTA-cG250) and had at least 1 post-baseline response assessment. The Evaluable Analysis Set includes 23 subjects who completed Cycle 1, 12 subjects who completed Cycle 2, and 4 subjects who completed Cycle 3.
Measure: Number; unit: participants
Arm/Group | Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 2 | 6
participants
  Cycle 1: Stable Disease | 2 | 2 | 5 | 2 | 2 | 6
  Cycle 1: Progressive Disease | 1 | 1 | 1 | 1 | 0 | 0
  Cycle 2: Partial Response | 0 | 0 | 1 | 0 | 0 | 0
  Cycle 2: Stable Disease | 1 | 1 | 2 | 1 | 0 | 2
  Cycle 2: Progressive Disease | 1 | 1 | 0 | 1 | 0 | 1
  Cycle 3: Stable Disease | 1 | 0 | 1 | 0 | 0 | 1
  Cycle 3: Progressive Disease | 0 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 1 year for each subject.
Description: AE documentation included onset/resolution dates, severity using NCI CTCAE (v3.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per subject at the maximum reported grade.
Groups:
- Total: 111-In-DOTA-cG250: On Day 1, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 5 mCi of 111-In.
  177-Lu-DOTA-cG250: On Day 8, 9, or 10, subjects received a single dose of 10 mg of cG250 coupled to DOTA and labeled with 30 to 70 mCi/m^2 of 177-Lu.
Arm/Group | Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 | Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250 | Total
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 1/6 | 0/3 | 1/3 | 2/8 | 6/26
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 3/3 | 2/3 | 6/8 | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 (N=3) | Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 (N=3) | Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 (N=6) | Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 (N=3) | Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 (N=3) | Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250 (N=8) | Total (N=26)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, 30 mCi/m^2 177-Lu-DOTA-cG250 (N=3) | Cohort 2, 40 mCi/m^2 177-Lu-DOTA-cG250 (N=3) | Cohort 3, 50 mCi/m^2 177-Lu-DOTA-cG250 (N=6) | Cohort 4, 60 mCi/m^2 177-Lu-DOTA-cG250 (N=3) | Cohort 5, 70 mCi/m^2 177-Lu-DOTA-cG250 (N=3) | Cohort 6, 65 mCi/m^2 177-Lu-DOTA-cG250 (N=8) | Total (N=26)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 0 | 1 | 5 | 11
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 1 | 4 | 8
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 3
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 3 | 2 | 5 | 16
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 3 | 6
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 3
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 2 | 5 | 3 | 1 | 3 | 15
Pyrexia (General disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 3
Malaise (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 4
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 3 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 3
Headache (Nervous system disorders) | 0 | 0 | 3 | 1 | 2 | 1 | 7
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 0 | 0 | 2 | 6
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less